CLINICAL TRIAL: NCT01716221
Title: An Objective Double-blind Evaluation of Bupropion and Citalopram in an Individual With Friedreich Ataxia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 11-1141
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Bupropion; Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Bupropion & Citalopram (Experimental): 100mg Bupropion & 20mg Citalopram taken orally one time per day or 100mg Bupropion & 10mg Citalopram taken orally one time per day or 50mg Bupropion & 20mg Citalopram taken orally one time per day 0r 50mg Bupropion & 10mg Citalopram taken orally one time per day
  Interventions: Drug: bupropion & Citalopram
- Bupropion & Placebo (Active Comparator): 100mg Bupropion & Placebo taken orally one time per day or 50mg Bupropion & Placebo taken orally one time per day
  Interventions: Drug: Bupropion & Placebo
- Placebo & Citalopram (Active Comparator): Placebo & 20mg Citalopram taken orally one time per day or Placebo & 10mg Citalopram taken orally one time per day
  Interventions: Drug: Placebo & Citalopram
- Placebo & Placebo (Placebo Comparator): Placebo & Placebo taken orally one time per day
  Interventions: Drug: Placebo & Placebo

INTERVENTIONS:
Drug: bupropion & Citalopram
  Arms: Bupropion & Citalopram
Drug: Bupropion & Placebo
  Arms: Bupropion & Placebo
Drug: Placebo & Citalopram
  Arms: Placebo & Citalopram
Drug: Placebo & Placebo
  Arms: Placebo & Placebo

SUMMARY:
The purpose of this study is to document the clinical effects of bupropion and citalopram in a single subject with Friedreich Ataxia.

DETAILED DESCRIPTION:
This is a double blind study with a single subject to objectively document the clinical effects of bupropion and citalopram in a single patient with Friedreich Ataxia (FA), whose disorder symptoms have improved with the use of these medications.

ELIGIBILITY:
Inclusion Criteria:

* Friedreich Ataxia

Exclusion Criteria:

* Unable to provide Informed Consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Klepitskaya, MD, Principal Investigator — University of Colorado, Denver

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participant: the participant received all intervention combinations in the following order: bupropion & Citalopram, then Bupropion & Placebo, then Placebo & Citalopram, then Placebo & Placebo
Period: Overall Study
Arm/Group | Study Participant
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Participant
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: International Cooperative Ataxia Rating Scale (ICARS)
Description: The ICARS is a 19 item rating scale of ataxia with the total score ranging from 0 to 100. A score of 0 means normal and higher scores represent worsened disease.
Time Frame: Assessements are performed in 5 different states in a single patient: baseline (Bupropion 100mg and Citalopram 20mg - unblinded), then blinded at 5 weeks (citalopram), 10 weeks (placebo), 15 weeks (bupropion), and 20 weeks (citalopram + bupropion)
Measure: Number; unit: units
Groups:
- Bupropion & Citalopram: 100mg Bupropion & 20mg Citalopram taken orally one time per day or 100mg Bupropion & 10mg Citalopram taken orally one time per day or 50mg Bupropion & 20mg Citalopram taken orally one time per day or 50mg Bupropion & 10mg Citalopram taken orally one time per day
  bupropion & Citalopram
- Bupropion & Placebo: 100mg Bupropion & Placebo taken orally one time per day or 50mg Bupropion & Placebo taken orally one time per day
  Bupropion & Placebo
- Placebo & Citalopram: Placebo & 20mg Citalopram taken orally one time per day or Placebo & 10mg Citalopram taken orally one time per day
  Placebo & Citalopram
- Placebo & Placebo: Placebo & Placebo taken orally one time per day
  Placebo & Placebo
- Baseline: unblinded 100mg Bupropion & 20mg Citalopram
Arm/Group | Bupropion & Citalopram | Bupropion & Placebo | Placebo & Citalopram | Placebo & Placebo | Baseline
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
units | 39 | 30 | 47 | 46 | 42

2. Primary Outcome: Friedreich Ataxia Rating Scale (FARS)
Description: A rating scale developed for Friedreich ataxia in evaluation of ataxia. Score range from 0-159 with a score of 0 meaning normal and greater scores indicating worsened disease.
Time Frame: Assessements are performed in 5 different states in a single patient: baseline (Bupropion 100mg and Citalopram 20mg - unblinded), then blinded at 5 weeks (citalopram), 10 weeks (placebo), 15 (bupropion), and 20 weeks (citalopram + bupropion)
Measure: Number; unit: points
Arm/Group | Baseline - Unblinded on Buproprion and Citalopram | Citalopram (Week 5) | OFF - Bupropion Placebo + Citalopram Placebo (Week 10) | Bupropion Only (Week 15) | Bupropion + Citalopram (Week 20)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
points | 43 | 41 | 47 | 42 | 45

3. Secondary Outcome: Comparison of FARS and ICARS
Description: Differences between FARS - ICARS at each treatment interval
Time Frame: as for outcome 2
Measure: Number; unit: points
Arm/Group | Baseline - Unblinded on Buproprion and Citalopram | Citalopram (Week 5) | OFF - Bupropion Placebo + Citalopram Placebo (Week 10) | Bupropion Only (Week 15) | Bupropion + Citalopram (Week 20)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
points | 1 | -6 | 1 | 12 | 6

4. Other Pre Specified Outcome: Hamilton Depression Rating Scale
Description: The Hamilton Depression Rating Scale is a 21 item questionnaire scored each item on a scale of 0 to 3 or 5. The max score is 66. Higher scores indicate worsened depression. All items are summed together to give a total score. A total score of 0-7 is considered normal, while total scores greater than 20 are indicative of moderate or greater depression.
Time Frame: as for outcome 2
Measure: Number; unit: units on a scale
Arm/Group | Baseline - Unblinded on Buproprion and Citalopram | Citalopram (Week 5) | OFF - Bupropion Placebo + Citalopram Placebo (Week 10) | Bupropion Only (Week 15) | Bupropion + Citalopram (Week 20)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
units on a scale | 7 | 10 | 2 | 3 | 4

ADVERSE EVENTS:
Groups:
- Bupropion & Citalopram: 100mg Bupropion & 20mg Citalopram taken orally one time per day or 100mg Bupropion & 10mg Citalopram taken orally one time per day or 50mg Bupropion & 20mg Citalopram taken orally one time per day 0r 50mg Bupropion & 10mg Citalopram taken orally one time per day
  bupropion & Citalopram
Arm/Group | Bupropion & Citalopram | Bupropion & Placebo | Placebo & Citalopram | Placebo & Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes